CLINICAL TRIAL: NCT02812134
Title: Impact of Oral Phosphorus Supplements on the 6-month Change in FGF23 Levels in Anorexic Adolescents Suffering From Undernutrition.
Acronym: IPSAASU
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Centre Hospitalier Universitaire, Amiens (Other)
Responsible Party: Sponsor
Other Study IDs: PI2015_843_0006
Record Dates: First submitted 2016-06-16; First posted 2016-06-24 (Estimated); Last update posted 2018-08-21 (Actual); Status verified 2018-08

CONDITIONS: Malnutrition
Keywords: phosphorus supplementation; FGF23; anorexic; adolescents; undernutrition
MeSH Terms: conditions — Malnutrition; Anorexia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- anorexic

SUMMARY:
Fibroblast growth factor 23 (FGF23) is a recently discovered phosphaturic hormone produced by osteocytes. It is involved in phosphate-calcium metabolism (via its phosphaturic action and inhibition of 1,25-OH vitamin D).

There are no published studies on the role of FGF23 in undernourished anorexic adolescents taking oral phosphorus supplements.

ELIGIBILITY:
Inclusion Criteria:

* Adolescents aged from 11 to 17
* Follow-up or hospitalisation for anorexia
* Overt undernutrition (clinical signs of undernutrition, body mass index and the Waterlow index)
* Social security coverage

Exclusion Criteria:

* Known pre-existing renal disorders
* Known constitutional disorders of phosphate-calcium metabolism
* Adult patients, legal guardianship, incarceration

Ages: 11 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: anorexic patients
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2015-06; Primary Completion 2018-08 (Estimated); Study Completion 2018-08 (Estimated)

PRIMARY OUTCOMES:
FGF23 | at inclusion and then once a month for 6 months.
  Change in the FGF23 level (U/ml) with regard to the exogenous phosphorus intake (doses of Phosphoneuros®, expressed in mg/kg/day)

CONTACTS AND LOCATIONS:
Overall Officials: Lydia LICHTENBERGER, PhD, Principal Investigator — CHU Amiens
Locations (1):
- CHU Amiens, Amiens, France